CLINICAL TRIAL: NCT00959608
Title: Modeling Effective Obesity Treatment to Reduce Disparities Through Primary Care
Brief Title: Think Health! A Personal Weight Management Program
Acronym: Think Health!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Shiriki K. Kumanyika, Ph.D., M.P.H./Professor of Epidemiology, University of Pennsylvania School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 804917
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Weight Management in adults; Reducing Health Disparities
MeSH Terms: conditions — Obesity | interventions — Alkalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basic (Active Comparator): Basic program participants receive 10-15 minute PCP weight management counseling at approximately four month intervals for up to 24 months and weight management materials.
  Interventions: Behavioral: Think Health! program
- Basic Plus (Experimental): Half of study participants are randomly assigned to Basic Plus program, where in addition to receiving the same intervention as the Basic program participants, the Basic Plus participants also receive counseling from a lifestyle coach at the primary care provider's office (monthly in year 1 and bimonthly in year 2).
  Interventions: Behavioral: Think Health! program; Behavioral: Basic Plus program

INTERVENTIONS:
Behavioral: Think Health! program — Brief 10-15 minute counseling with Primary Care Provider for weight management, Participant binder with eating, physical activity and stress management educational materials, adapted from the Diabetes Prevention Program (DPP)(Knowler et al, 2002; DPP Research Group, 2002), physical activity resource guide, and telephonic health related messages (year 2).
Behavioral: Basic Plus program — 15 minute counseling sessions with lifestyle coach, in addition to the Basic Think Health! program intervention.
  Arms: Basic Plus

SUMMARY:
Think Health! A Personal Weight Management Program, or "¡Vive Saludable! Un programa personalizado de control de peso" aims to improve the treatment of obesity in adults in the general population, by conducting research with men and women recruited from primary care medical practices. The study has a particular focus on African Americans and Latino. The design is randomized trial of the effectiveness of two versions of a lifestyle weight loss program called delivered by primary care providers (PCP) and ancillary staff at 5 clinical practice sites to their own patients. The two versions of the lifestyle weight loss program are called Basic (minimal counseling provided by PCP every four months) and Basic Plus (same PCP counseling plus additional counseling by specially trained ancillary practice staff acting as Lifestyle Coaches (LC), monthly for the first 12 months and then every other month for up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

1. Women and men
2. Ages 18 to 70 years
3. Body mass index > 25 kg/m2 but < 55 kg/m2 or who weigh <400 pounds.

Exclusion Criteria:

1. Pregnancy or lactation, since contraindicated for weight loss or affecting weight status
2. Weight loss > 10 pounds in the previous 3 months
3. Current use of weight loss medications
4. Use of medications known to result in significant weight gain (e.g., oral steroids or second generation anti-psychotics)
5. Psychiatric disorders including untreated major depression, psychosis, bulimia nervosa, and substance abuse
6. Active chemo- or radiation therapy
7. Unstable renal, hepatic, or cardiovascular disease, including malignant arrhythmias
8. Recent (past 3 months) history of myocardial infarction, stroke, or congestive heart failure
9. Participants age < 18 will be excluded because we are only using adult practices and a different type of program would be needed for patients < 18, and age > 70 years will be excluded because our experience has been that a specially tailored program would be needed. As a design consideration, we wanted to decrease the heterogeneity of the program.
10. Participants with a BMI > 55 kg/m2 will be excluded because they are likely to require more extensive medical and behavioral care than can be provided in this study.
11. More than 1 participant residing in the same household will be excluded to avoid contamination across the treatment conditions.
12. Final exclusion criteria will be determined in collaboration with participating primary care providers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight, as measured at months 0, 12, 24 (or at final visit). | Up to 24 months

SECONDARY OUTCOMES:
Blood pressure, height, and waist measurements; surveys to assess health behavior changes; and attendance at treatment visits. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiriki K Kumanyika, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (5):
  - Penn Family Care at St. Leonard's Court, Philadelphia, Pennsylvania
  - PennCare- Edward S. Cooper Practice of General Internal Medicine, Philadelphia, Pennsylvania
  - Greenhouse Internists, Philadelphia, Pennsylvania
  - Einstein Community Health Associates, Philadelphia, Pennsylvania
  - Northeast Family Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Kumanyika SK, Morales KH, Allison KC, Russell Localio A, Sarwer DB, Phipps E, Fassbender JE, Tsai AG, Wadden TA. Two-Year Results of Think Health! inverted exclamation markVive Saludable!: A Primary Care Weight-Management Trial. Obesity (Silver Spring). 2018 Sep;26(9):1412-1421. doi: 10.1002/oby.22258. Epub 2018 Aug 29. PMID 30160061